CLINICAL TRIAL: NCT06301581
Title: Retrospective Analysis of Speech Performance Using the HiRes Ultra and HiRes Ultra 3D Cochlear Implant
Status: Recruiting | Type: Observational
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ABIntl-23-42
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: HiRes Ultra or HiRes Ultra 3D Version V2 newly implanted on this side
- Group 2: HiRes Ultra or HiRes Ultra 3D Version V2 implanted following an Ultra Version V1 device failure on the same ear

SUMMARY:
This is a retrospective study designed to collect speech perception results for HiRes Ultra CI and HiRes Ultra 3D CI users as measured in the clinical routine and to confirm the performance of these devices.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral HiRes Ultra CI or HiRes Ultra 3D CI users including

  * Ultra Version V2 newly implanted on this side (Group 1)
  * Ultra Version V2 users implanted following an Ultra Version V1 device failure in the same ear (Group 2)
* Informed consent signed

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The studied population consists of all CI users implanted with a HiRes Ultra Version V2 or HiRes Ultra 3D Version V2 CI at the Medical University of Hannover in Germany (MHH).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Freiburger monosyllabic word recognition score in quiet in the implanted ear | 12 months after device activation
  Score obtained with the Freiburger Monosyllabic word test

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Büchner, Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany